CLINICAL TRIAL: NCT03140423
Title: Cluster-randomized Non-inferiority Trial Comparing Mupirocin vs Iodophor for Nasal Decolonization of ICU Patients to Assess Impact on S. Aureus Clinical Cultures and All-cause Bloodstream Infection During Routine Chlorhexidine Bathing
Brief Title: Mupirocin-Iodophor ICU Decolonization Swap Out Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Hospital Corporation of America (Industry); University of California, Irvine (Other); University of Massachusetts, Amherst (Other); Rush University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Platt, Professor and Department Chair, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PH000599A
Record Dates: First submitted 2017-04-12; First posted 2017-05-04 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Staphylococcus Aureus
Keywords: MRSA; healthcare-associated infections; mupirocin; iodophor; resistance
MeSH Terms: conditions — Staphylococcal Infections; Cross Infection

STUDY DESIGN:
Intervention Model Description: Non-inferiority cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Routine Care (Mupirocin/CHG) (Active Comparator): ICU nasal decolonization with mupirocin twice daily for 5 days in the context of chlorhexidine for daily bathing
  Interventions: Drug: Arm 1. Routine Care (Mupirocin/CHG)
- Arm 2: Iodophor/CHG Decolonization (Active Comparator): ICU nasal decolonization with iodophor twice daily for 5 days in the context of chlorhexidine for daily bathing
  Interventions: Drug: Arm 2. Iodophor/CHG Decolonization

INTERVENTIONS:
Drug: Arm 1. Routine Care (Mupirocin/CHG) — The intervention / decolonization regimen will consist of 5 days of topical intranasal mupirocin ointment (bilateral nares, twice daily) on ICU admission, in the context of continued daily baths with 2% chlorhexidine cloths.
  Arms: Arm 1: Routine Care (Mupirocin/CHG)
Drug: Arm 2. Iodophor/CHG Decolonization — The intervention / decolonization regimen will consist of 5 days of topical intranasal iodophor (10% povidone-iodine nasal swabs) (bilateral nares, twice daily) on ICU admission, in the context of continued daily baths with 2% chlorhexidine cloths.
  Arms: Arm 2: Iodophor/CHG Decolonization

SUMMARY:
The Swap Out Trial is a cluster randomized controlled trial of HCA hospitals, evaluating the non-inferiority of two decolonization regimens:

Arm 1 Routine Care: ICU nasal decolonization with mupirocin twice daily for 5 days in the context of chlorhexidine for daily bathing; Arm 2 Intervention: ICU nasal decolonization with iodophor twice daily for 5 days in the context of chlorhexidine for daily bathing Note: that enrolled "subjects" represents 137 individual HCA Hospitals (representing ~235 ICUs) that have been randomized.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria includes all U.S. HCA hospitals with an adult ICU;
* Note: Unit of randomization is the hospital, but the participants are hospital adult ICUs
* All patients within adult ICUs are included, including rare patients <18 years and >=12 years.

Exclusion Criteria:

* Exclusion criteria includes ICUs with an average length of stay of less than 2 days;
* HCA hospitals that are not able to transfer or merge data into the centralized data warehouse for the baseline and intervention periods of the study are also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 353323 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Platt, MD, MS, Principal Investigator — Harvard Pilgrim Health Care Institute; Susan Huang, MD, MPH, Study Director — University of California, Irvine
Locations (137):
- United States (137):
  - Riverside Community Hospital, Riverside, California
  - Regional Medical Center of San Jose, San Jose, California
  - Good Samaritan Hospital, San Jose, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - West Hills Hospital & Medical Center, West Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Swedish Medical Center, Denver, Colorado
  - Sky Ridge Medical Center, Denver, Colorado
  - Presbyterian St. Luke's Medical Center, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - North Suburban Medical Center - JV, Thornton, Colorado
  - JFK Medical Center, Atlantis, Florida
  - Aventura Hospital, Aventura, Florida
  - Blake Medical Center, Bradenton, Florida
  - Brandon Regional, Brandon, Florida
  - Oak Hill Hospital, Brooksville, Florida
  - Englewood Community Hospital, Englewood, Florida
  - Fort Walton Medical Center, Fort Walton Beach, Florida
  - Lawnwood Regional Medical Center, Ft. Pierce, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Regional Medical Center Bayonet Point, Hudson, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Poinciana Medical Center, Kissimmee, Florida
  - Lake City Medical Center, Lake City, Florida
  - Largo Medical Center, Largo, Florida
  - Palms West Hospital, Loxahatchee Groves, Florida
  - Northwest Medical Center, Margate, Florida
  - Mercy Hospital, Miami, Florida
  - Kendall Regional Medical Center, Miami, Florida
  - Twin Cities Hospital, Niceville, Florida
  - Ocala Regional Medical Center, Ocala, Florida
  - West Marion Community Hospital, Ocala, Florida
  - Raulerson Hospital, Okeechobee, Florida
  - Orange Park Medical Center, Orange Park, Florida
  - Gulf Coast Medical Center, Panama City, Florida
  - West Florida Hospital, Pensacola, Florida
  - Plantation General Hospital, Plantation, Florida
  - Westside Regional Medical Center, Plantation, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - St. Lucie Medical Center, Port Saint Lucie, Florida
  - Central Florida Regional Hospital, Sanford, Florida
  - Doctor's Hospital Sarasota, Sarasota, Florida
  - Northside Hospital, St. Petersburg, Florida
  - St. Petersburg General Hospital, St. Petersburg, Florida
  - South Bay Hospital, Sun City Center, Florida
  - Capital Regional Medical Center, Tallahassee, Florida
  - University Hospital & Medical Center, Tamarac, Florida
  - Medical Center of Trinity, Trinity, Florida
  - JFK Medical Center - North Campus, West Palm Beach, Florida
  - Doctor's Hospital Augusta, Augusta, Georgia
  - Cartersville Medical Center, Cartersville, Georgia
  - Fairview Park, Dublin, Georgia
  - Coliseum Medical Centers - Main, Macon, Georgia
  - Coliseum Medical Centers - Northside, Macon, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Eastside Medical Center, Snellville, Georgia
  - West Valley Medical Center, Caldwell, Idaho
  - Eastern Idaho Regional, Idaho Falls, Idaho
  - Terre Haute Regional Hospital, Terre Haute, Indiana
  - Menorah Medical Center, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wesley Woodlawn Hospital, Wichita, Kansas
  - Greenview Regional Hospital, Bowling Green, Kentucky
  - Rapides Regional Medical Center, Alexandria, Louisiana
  - Lakeview Regional Medical Center, Covington, Louisiana
  - Tulane University Hospital & Clinic, New Orleans, Louisiana
  - Garden Park Medical Center, Gulfport, Mississippi
  - Belton Regional Medical Center, Belton, Missouri
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Lee's Summit Medical Center, Lee's Summit, Missouri
  - Sunrise Hospital & Medical Center, Las Vegas, Nevada
  - Mountainview Hospital - Vegas, Las Vegas, Nevada
  - Southern Hills Hospital - Vegas, Las Vegas, Nevada
  - Parkland Medical Center, Derry, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Spotsylvania Regional Medical Center, Fredericksburg, Pennsylvania
  - Trident Regional Medical Center, Charleston, South Carolina
  - Grand Strand Regional Medical Center, Myrtle Beach, South Carolina
  - Summerville Medical Center, Summerville, South Carolina
  - Colleton Medical Center, Walterboro, South Carolina
  - Parkridge Medical Center, Chattanooga, Tennessee
  - Parkridge East Hospital, Chattanooga, Tennessee
  - Hendersonville Medical Center, Hendersonville, Tennessee
  - Summit Medical Center, Hermitage, Tennessee
  - Stonecrest Medical Center, Nashville, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Skyline Medical Center, Nashville, Tennessee
  - Southern Hills Medical Center, Nashville, Tennessee
  - Medical Center of Arlington, Arlington, Texas
  - South Austin Hospital, Austin, Texas
  - North Austin Medical Center, Austin, Texas
  - Valley Regional Medical Center, Brownsville, Texas
  - Conroe Regional Medical Center, Conroe, Texas
  - Corpus Christi Medical Center - Doctor's, Corpus Christi, Texas
  - Corpus Christi Medical Center - The Heart Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Denton Regional Medical Center, Denton, Texas
  - Las Palmas Medical Center, El Paso, Texas
  - Del Sol Medical Center, El Paso, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - East Houston Regional Medical Center, Houston, Texas
  - West Houston Medical Center, Houston, Texas
  - Las Colinas Medical Center, Irving, Texas
  - Kingwood Medical Center, Kingwood, Texas
  - Medical Center of Lewisville, Lewisville, Texas
  - Rio Grande Regional Hospital, McAllen, Texas
  - Medical Center of McKinney, McKinney, Texas
  - North Hills Hospital, North Richland Hills, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - Medical Center of Plano, Plano, Texas
  - Round Rock Hospital, Round Rock, Texas
  - Metropolitan Methodist Hospital, San Antonio, Texas
  - Methodist Hospital, San Antonio, Texas
  - Methodist Specialty & Transplant Hospital, San Antonio, Texas
  - Methodist Stone Oak Hospital, San Antonio, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Northeast Methodist Hospital, San Antonio, Texas
  - Mainland Medical Center, Texas City, Texas
  - Clearlake Regional Medical Center, Webster, Texas
  - Lakeview Hospital, Bountiful, Utah
  - Ogden Regional Medical Center, Ogden, Utah
  - Timpanogos Regional Medical Center, Orem, Utah
  - Mountain View Hospital - Utah, Payson, Utah
  - LewisGale Hospital - Montgomery, Blacksburg, Virginia
  - John Randolph Medical Center, Hopewell, Virginia
  - LewisGale Hospital - Alleghany, Low Moor, Virginia
  - LewisGale Hospital - Pulaski, Pulaski, Virginia
  - Reston Hospital, Reston, Virginia
  - Henrico Doctors' Hospital - Retreat Campus, Richmond, Virginia
  - CJW Medical Center (Chippenham Campus), Richmond, Virginia
  - CJW Medical Center (Johnston Willis Campus), Richmond, Virginia
  - Henrico Doctors' Hospital - Forest Campus, Richmond, Virginia
  - Henrico Doctors' Hospital - Parham Campus, Richmond, Virginia
  - LewisGale Medical Center, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang SS, Septimus EJ, Kleinman K, Heim LT, Moody JA, Avery TR, McLean L, Rashid S, Haffenreffer K, Shimelman L, Staub-Juergens W, Spencer-Smith C, Sljivo S, Rosen E, Poland RE, Coady MH, Lee CH, Blanchard EJ, Reddish K, Hayden MK, Weinstein RA, Carver B, Smith K, Hickok J, Lolans K, Khan N, Sturdevant SG, Reddy SC, Jernigan JA, Sands KE, Perlin JB, Platt R. Nasal Iodophor Antiseptic vs Nasal Mupirocin Antibiotic in the Setting of Chlorhexidine Bathing to Prevent Infections in Adult ICUs: A Randomized Clinical Trial. JAMA. 2023 Oct 10;330(14):1337-1347. doi: 10.1001/jama.2023.17219. PMID 37815567
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38639723/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 137 out of 178 HCA Healthcare hospitals were recruited for this trial of adult ICUs. There was an 18-month intervention period from November 1, 2017 through April 30, 2019.
Pre-assignment Details: 353,323 patients were involved in the intervention period among adult ICUs from the 137 participating hospitals.
Units Other Than Participants: Hospitals
Period: Overall Study
Arm/Group | Arm 1: Routine Care (Mupirocin/CHG) | Arm 2: Iodophor/CHG Decolonization
Started | 168301; 68 Hospitals | 185022; 69 Hospitals
Completed | 168301; 66 Hospitals | 185022; 68 Hospitals
Not Completed | 0; 2 Hospitals | 0; 1 Hospitals

BASELINE CHARACTERISTICS:
Population: Number of Participant totals reflect total Intervention participants. 137 hospitals were randomized to a study group, 69 began the assigned intervention. 1 hospital withdrew from the intervention arm and 2 hospitals withdrew from the control arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Routine Care (Mupirocin/CHG) | Arm 2: Iodophor/CHG Decolonization | Total
Number analyzed (Participants) | 168301 | 185022 | 353323
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Overall number of participants reflect participants during the Intervention period.
  years
    Age | 66.0 [54.0 to 76.0] | 66.0 [54.0 to 76.0] | 66.0 [53.0 to 76.0]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Proportion of female study participants during intervention study phase. Population: Small differences in the number of patients with various characteristics reflect missing data in the electronic health record.
  Participants
    Sex: number analyzed (Participants) | 168219 | 184950 | 353169
    Sex: Female | 78074 | 85194 | 163268
    Sex: Male | 90145 | 99756 | 189901
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Small differences in the number of patients with various characteristics reflect missing data in the electronic health record.
  Participants
    Race: number analyzed (Participants) | 155666 | 171982 | 327648
    Race: Black or African American | 21901 | 27776 | 49677
    Race: White | 126749 | 135060 | 261809
    Race: Other | 7016 | 9146 | 16162

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ICU-attributable Staphylococcus Aureus Clinical Cultures
Description: Methicillin-resistant Staphylococcus aureus (MRSA) and Methicillin-susceptible Staphylococcus aureus (MSSA) clinical cultures attributable to participating ICUs. Defined as occurring >2 days into a participating ICU stay through 2 days following ICU discharge. NOTE: this outcome is intended for the primary manuscript.
Time Frame: 18-month intervention
Population: The total number of participants analyzed reported here is from the intervention period.
Measure: Number; unit: participants
Arm/Group | Arm 1: Routine Care (Mupirocin/CHG) | Arm 2: Iodophor/CHG Decolonization
Number analyzed (Participants) | 168301 | 185022
participants | 2708 | 3563

2. Secondary Outcome: Number of Participants With ICU Attributable MRSA Clinical Cultures
Description: Methicillin-resistant Staphylococcus aureus (MRSA) clinical cultures attributable to participating ICUs. Defined as occurring >2 days into a participating ICU stay through 2 days following ICU discharge. NOTE: this outcome is intended for the primary manuscript.
Time Frame: 18-month intervention
Population: The total number of participants analyzed reported here is from the intervention period.
Measure: Number; unit: participants
Arm/Group | Arm 1: Routine Care (Mupirocin/CHG) | Arm 2: Iodophor/CHG Decolonization
Number analyzed (Participants) | 168301 | 185022
participants | 1377 | 1682

3. Secondary Outcome: Number of Participants With ICU-attributable Bloodstream Infections
Description: All-cause bloodstream infection attributable to participating ICUs. Defined as occurring >2 days into a participating ICU stay through 2 days following ICU discharge.Includes subsets of gram positive (GP), gram negative (GN) and fungal (candida) bloodstream infections, as well as key pathogens such as S. aureus (MRSA and MSSA). NOTE: this outcome is intended for the primary manuscript.
Time Frame: 18-month intervention
Population: The total number of participants analyzed reported here is from the intervention period.
Measure: Number; unit: participants
Arm/Group | Arm 1: Routine Care (Mupirocin/CHG) | Arm 2: Iodophor/CHG Decolonization
Number analyzed (Participants) | 168301 | 185022
participants | 1766 | 1956

ADVERSE EVENTS:
Time Frame: 18 Months
Description: There were 2 adverse events, both in the Iodophor-CHG group. One involved mild nasal pruritus, and one involved total body hives requiring treatment. Both resolved on discontinuation of decolonization.
Arm/Group | Arm 1: Routine Care (Mupirocin/CHG) | Arm 2: Iodophor/CHG Decolonization
All-Cause Mortality (participants affected / at risk) | 0/168301 | 0/185022
Serious Adverse Events (participants affected / at risk) | 0/168301 | 0/185022
Other Adverse Events (participants affected / at risk) | 0/168301 | 2/185022
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Routine Care (Mupirocin/CHG) (N=168301) | Arm 2: Iodophor/CHG Decolonization (N=185022)
Other (Not Including Serious) Adverse Event (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT03140423/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT03140423/SAP_001.pdf